CLINICAL TRIAL: NCT03158298
Title: Association of Schistosomiasis Seropositivity With Adverse Birth Events in Migrants From Bilharzia-endemic Areas
Brief Title: Seropositivity and Adverse Birth Events in Migrants From Bilharzia-endemic Areas
Acronym: Bilharzia
Status: Terminated | Type: Observational
Why Stopped: due to lack of recruitment
Sponsor: Jena University Hospital (Other)
Collaborators: Technical University of Munich (Other); Charite University, Berlin, Germany (Other); University Hospital in Halle (Other)
Responsible Party: Sponsor
Other Study IDs: ZKS0094
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Schistosomiasis
MeSH Terms: conditions — Schistosomiasis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Placenta (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Specimen collection — Maternal blood sample of 10 ml collected by venepuncture upon delivery

SUMMARY:
The study intends to examine the association between schistosomiasis seropositivity and adverse pregnancy outcomes.

It aims at the verification of the hypothesis that in pregnant women originating from endemic areas for schistosomiasis, positive serology is associated with reduced Infant birth weight.

DETAILED DESCRIPTION:
Schistosomiasis is a widespread helminthic infection, with an estimated 249 million people in 78 countries requiring preventive treatment each year. This infection has a significant association with morbidity worldwide. Earlier studies performed in endemic Areas showed that the reproductive tract was affected in more than 60% of the women who excreted S. haematobium ova in urine. Transplacental transmission has not been observed, but schistosomiasis of the pregnant uterus has been reported and placental schistosomiasis has been associated with stillbirth. Placental schistosomiasis (i.e. detection of schistosomiasis eggs in placental tissue) has been reported occasionally. Schistosomiasis has been postulated to be associated with premature delivery and low birth weight; however, existing data are inconsistent.

Migration to the European Union was estimated at 1.7 million people in 2012. Migrants were predominantly from Africa and Asia. In these areas schistosomiasis has an estimated prevalence of 10-20%. While a large number of migrants from schistosomiasis-endemic areas enter Europe and receive Access to health care, many of them are unaware of helminthic infections they may have been exposed to, and their potential outcomes.

Treatment of schistosomiasis during pregnancy is a matter of debate. The German society for tropical medicine recommends treatment with praziquantel only after the completion of pregnancy. Conversely, the South African Medicines Formulary suggests that pregnant women should be offered treatment individually and that they should not necessarily be excluded during treatment campaigns. By quantifying the effects of Schistosoma infection on pregnancy outcomes this study will help clinicians in deciding on the question of treatment during pregnancy.

The aim of the study is to examine the association of maternal schistosomiasis on adverse birth outcomes (as defined by low birth weight, premature delivery or stillbirth) in migrants to Europe from schistosomiasis endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Immigration from a country/geographic area with declared endemic schistosomiasis according to World Health Organization criteria
* Signed informed consent

Exclusion Criteria:

* Placenta pathology of any cause
* Any medical condition affecting fetal growth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study objectives pertain to pregnant women
Study Population: Pregnant women aged above 18, who migrated to Europe from geographic regions with endemic schistosomiasis
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Schleenvoigt, M.D., Principal Investigator — Center for Infectious Diseases and Infection Control, Jena University Hospital
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Pregnant women >18 years originally from endemic countries and areas for Bilharzia (as defined by WHO) who give written informed consent to the study.
Period: Overall Study
Arm/Group | Study Group
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — refers on the gender of newborns (82 pregnancies with 82 mothers and 82 newborns)
  Participants
    Female | 30
    Male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 82
Schistosomiasis Serology [Number; unit: participants] | 82
gestational age [Median (Standard Deviation); unit: weeks] | 39.71 (2.43)
birth weight [Median (Standard Deviation); unit: g] | 3318 (623)

OUTCOME MEASURES:

1. Primary Outcome: Schistosoma Serology
Description: Presence of Schistosoma antibodies in maternal serum
Time Frame: 6 month after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 82
Participants | 0

2. Secondary Outcome: Birth Weight
Description: Infant birth weight
Time Frame: 1 hour upon delivery
Measure: Mean (Standard Deviation); unit: gramm
Arm/Group | Study Group
Number analyzed (Participants) | 82
gramm | 3273 (573)

3. Secondary Outcome: Preterm Birth
Description: Onset of delivery at a gestational age below 37 weeks
Time Frame: 24 hours before delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 82
Participants | 5

4. Secondary Outcome: Intrauterine Growth Restriction
Description: Fetal weight below the 10th percentile for the estimated gestational age
Time Frame: 48 hours after delivery
Population: all
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 82
Participants | 7

5. Secondary Outcome: Stillbirth
Description: Fetus delivered without signs of life at gestational age between 20 and 28 weeks
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 82
Participants | 0

ADVERSE EVENTS:
Time Frame: adverse event data collection was not applicable to our study
Description: adverse event data collection was not applicable to our observational study
Groups:
- Study Group: 82 mother-child pairs; women initially migrated from Bilharzia endemic countries
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03158298/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT03158298/ICF_001.pdf